CLINICAL TRIAL: NCT06621043
Title: Assessing the Safety and Efficacy of Full-Spectrum Medicinal Cannabis Plant Extract 0.08% THC (NTI164) in the Treatment of Rett Syndrome (RTT)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fenix Innovation Group (Industry)
Collaborators: Neurotech International Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTIRTT1
Record Dates: First submitted 2024-09-11; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Rett Syndrome
Keywords: RTT
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active NTI164 Arm (Experimental): Participants in this arm receive Full-Spectrum Medicinal Cannabis Plant Extract containing 0.08% THC (NTI164), targeted at treating symptoms of Rett syndrome (RTT) in children and young people. The intervention starts with a daily initial dose of 5 mg/kg, which is increased gradually over a four-week up-titration phase to a maximum of 20 mg/kg per day, depending on individual tolerance. Participants then continue at their maximum tolerated dose for eight weeks during the treatment phase. The study concludes with a four-week down-titration phase, where the dosage is reduced by 5 mg/kg each week. The effectiveness of the treatment is monitored through specialized questionnaires and full blood examinations throughout the study duration.
  Interventions: Drug: NTI164

INTERVENTIONS:
Drug: NTI164 — Full-Spectrum Medicinal Cannabis Plant Extract containing 0.08% THC, administered orally starting with a dose of 5 mg/kg, titrated up to 20 mg/kg based on tolerance, followed by a maintenance phase at the maximum tolerated dose, and concluding with a gradual dose reduction.

SUMMARY:
This 18-week open-label study examines the effectiveness of Full-Spectrum Medicinal Cannabis Plant Extract containing 0.08% THC (NTI164) in treating Rett syndrome (RTT) in children and young people. The study aims to determine the impact of NTI164 on RTT symptoms over a 16-week treatment period.

Participants will start with a daily dose of 5 mg/kg of NTI164, which will be gradually increased over four weeks until they reach either the maximum tolerated dose or 20 mg/kg per day. They will then maintain this dose for eight weeks. Following this treatment phase, the dosage will be reduced by 5 mg/kg each week for four weeks until treatment concludes.

The effectiveness of the treatment will be assessed using tailored questionnaires that measure changes in the patients' conditions. Additionally, full blood examinations will be conducted at multiple points throughout the study to monitor the effects of the treatment.

DETAILED DESCRIPTION:
This study is an 18-week open-label trial designed to assess the effectiveness of Full-Spectrum Medicinal Cannabis Plant Extract containing 0.08% THC (NTI164) on the severity of symptoms in children and young people with Rett syndrome (RTT). The main objective is to determine how well NTI164 alleviates the symptoms of RTT over a 16-week treatment period.

The study involves multiple phases:

1. **Up-titration Phase (4 weeks):** Treatment begins with an initial daily dose of 5 mg/kg of NTI164. Over the first four weeks, this dose is incrementally increased based on patient tolerance, aiming for a maximum daily dose of 20 mg/kg.
2. **Treatment Phase (8 weeks):** Once the maximum tolerated dose is established, participants continue to receive this dose for the following eight weeks. This phase focuses on maintaining a steady dosage to observe the therapeutic effects on RTT symptoms.
3. **Down-titration Phase (4 weeks):** After completing the treatment phase, the dosage is systematically reduced by 5 mg/kg each week for four weeks until treatment cessation. This gradual reduction helps in assessing any withdrawal effects and the stability of symptom improvement post-treatment.

Throughout the study, the efficacy of NTI164 is evaluated using specifically designed questionnaires that track changes in the emotional, behavioral, and cognitive functions of the participants, providing insights into how the treatment impacts various aspects of RTT. Additionally, full blood examinations are conducted at key points during the study to monitor the physiological responses to the treatment and to ensure the safety and tolerability of NTI164. This comprehensive approach allows for a detailed assessment of both the immediate and longer-term effects of the medicinal cannabis extract on Rett syndrome symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Girls and women, aged 5-20 years
* Weight greater than or equal to 12kg
* Classical/typical RTT
* Documented disease-causing mutation in MECP2 gene
* At least 6 months post regression at screening (ie. no loss or degradation in ambulation, hand function, speech, nonverbal communicative or social skills within 6 months of screening) Rett Syndrome Clinical Severity Scale rating of 10-36
* CGI score of 4 or higher.
* Stable pattern of seizures, or has had no seizures, within 8 weeks of screening.

Exclusion Criteria:

* Current clinically significant cardiovascular, endocrine (such as hypo- or hyperthyroidism, type 1 diabetes, or uncontrolled type 2 diabetes), renal, hepatic, respiratory, or gastrointestinal disease (such as celiac disease or inflammatory bowel disease), or major surgery planned during the study.
* Known history or symptoms of long QT syndrome.
* QTcF interval >450 ms, history of risk factor for torsades de pointes or clinically significant QT prolongation deemed to increase risk.
* Treatment with insulin, IGF-1, or growth hormone within 12 weeks of baseline.
* Currently receiving treatment with DAYBUETM (trofinetide).
* Currently using other unregistered drugs for the treatment of Rett syndrome such as Anavex.
* Currently using or has used recreational or medicinal cannabis, cannabinoid-based medications (including Sativex®, or Epidiolex®) within the 12 weeks prior to screening and is unwilling to abstain for the duration of the trial.
* Participant has any known or suspected hypersensitivity to cannabinoids or any of the excipients.

Ages: 5 Years to 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 14 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rett Syndrome: Symptom Index Score | Baseline (pre-dose), 4, 12, 16 weeks post-commencement of treatment
  The Rett Syndrome: Symptom Index Score (RTT: SIS) measures the severity of various symptoms in individuals with Rett syndrome. Individual scores are from 0 to 7 with lower scores reflecting improvement or milder symptoms.

SECONDARY OUTCOMES:
Clinical Global Impression - Improvement (CGI-I) | Baseline (pre-dose), 4, 12, 16 weeks post-commencement of treatment
  The CGI-I (Clinical Global Impressions - Improvement) scale rates patient improvement on a scale from 1 to 7. Lower scores indicate better improvement.
Rett Syndrome Behaviour Questionnaire | Baseline (pre-dose), 4, 12, 16 weeks post-commencement of treatment.
  The Rett Syndrome Behaviour Questionnaire (RSBQ) assesses behavioural symptoms in individuals with Rett syndrome. Individual items are scored from 0 to 2. Higher total scores indicate more severe behavioural issues, meaning lower scores reflect better behavioural functioning.
RTT-Clinician Domain Specific Concerns - Visual Analog Scale | Baseline (pre-dose), 4, 12, 16 weeks post-commencement of treatment.
  The Rett Syndrome Clinician Domain Specific Concerns Visual Analog Scale (RTT-DSC-VAS) assesses clinician concerns across specific domains of Rett syndrome. Each domain is scored on a scale from 0 to 7, with higher scores reflecting greater impairment in specific areas, while lower scores suggest less concern.
Communication and Symbolic Behaviour Scales Developmental Profile™ Infant-Toddler Checklist | Baseline (pre-dose), 4, 12, 16 weeks post-commencement of treatment.
  The Communication and Symbolic Behavior Scales Developmental Profile Infant-Toddler Social Composite (CSBS-DP-IT Social) assesses early social communication skills in young children. Individual items are scored on a scale from 0 to 2, with higher scores indicating stronger social communication abilities. A lower total score reflects more social communication difficulties, while a higher score suggests better social engagement and communication skills.
Impact of Childhood Neurological Disability Scale | Baseline (pre-dose), 4, 12, 16 weeks post-commencement of treatment.
  The Impact of Childhood Neurological Disability Scale (ICND) assesses the impact of neurological disabilities on a child's daily life and functioning. Each item is scored from 0 to 3, where higher scores indicate greater disability impact. A lower total score reflects less impact or better functioning, while higher scores suggest more significant limitations due to the neurological condition.
Rett Syndrome Caregiver Burden Inventory | Baseline (pre-dose), 4, 12, 16 weeks post-commencement of treatment.
  The Rett Syndrome Caregiver Burden Inventory (RTT CBI) measures the burden experienced by caregivers of individuals with Rett syndrome. Individual items are scored from 0 to 4, with higher scores indicating a greater caregiver burden. Lower scores reflect less burden or stress, while higher scores suggest increased strain and challenges for caregivers.
The Overall Quality of Life Rating of the Impact of Childhood Neurological Disability Scale | Baseline (pre-dose), 4, 12, 16 weeks post-commencement of treatment.
  The Overall Quality of Life Rating of the Impact of Childhood Neurological Disability Scale (ICND-QoL) is completed by the caregiver, who rates the child's overall quality of life on a scale from 0 to 6, with 0 indicating the worst possible quality of life and 6 indicating the best. Higher scores reflect a more positive perception of the child's quality of life, while lower scores suggest a greater negative impact of the neurological condition.

CONTACTS AND LOCATIONS:
Locations (1):
- The Childrens Hospital at Westmead, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared as per commercial in confidence restrictions.